CLINICAL TRIAL: NCT00146133
Title: Effect of Weight Loss and Physical Training on Musculoskeletal Status, Physical Function, and Quality-of-Life in Physically Limited, Obese, Elderly Subjects
Brief Title: Weight Loss and Exercise in Physically Limited Obese Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KO7AG2116401; KO7AG2116401
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2005-09

CONDITIONS: Obesity; Frailty; Elderly
Keywords: Obesity, Aging, Frailty, exercise, weight loss
MeSH Terms: conditions — Obesity; Frailty; Motor Activity; Weight Loss | interventions — Diet; Exercise

INTERVENTIONS:
Behavioral: diet, exercise

SUMMARY:
The overall purpose of this research is to determine the effect of weight loss and physical training on quality of life, physical function, metabolism, bone strength, body fat and muscle mass.

DETAILED DESCRIPTION:
Obesity causes serious medical complications and impairs quality of life. Moreover, in elderly persons, obesity can lead to frailty because of decreased strength, joint function, balance and mobility associated with aging. The primary objective of this study is to evaluate the effect of weight loss and physical training on physical function, body composition, metabolism and quality of life in frail, obese elderly men and women. Subjects are randomized to either control or 10% weight loss plus physical training.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI 30 or greater) elderly (age 65 years or older) Frailty

Exclusion Criteria:

* Major chronic disease or any condition that would interfere with exercise or dietary restriction, in which exercise or dietary restriction are contraindicated, or that would interfere with interpretation of results. Examples include cardiopulmonary disease, unstable disease, severe orthopedic or neuromuscular impairments, dementia, history of malignancy during the past 5 yr, current use of bone acting drugs.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28
Dates: Start 2003-01; Study Completion 2004-12

PRIMARY OUTCOMES:
physical function and body composition

SECONDARY OUTCOMES:
quality of life, metabolic markers

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Villareal DT, Banks M, Siener C, Sinacore DR, Klein S. Physical frailty and body composition in obese elderly men and women. Obes Res. 2004 Jun;12(6):913-20. doi: 10.1038/oby.2004.111. PMID 15229329
- [Result] Villareal DT, Banks M, Sinacore DR, Siener C, Klein S. Effect of weight loss and exercise on frailty in obese older adults. Arch Intern Med. 2006 Apr 24;166(8):860-6. doi: 10.1001/archinte.166.8.860. PMID 16636211